CLINICAL TRIAL: NCT01615861
Title: Evaluation of Clinical Outcomes Following Implantation of a Sub-2mm Hydrophilic MICS Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 714
Record Dates: First submitted 2012-05-29; First posted 2012-06-11 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IOL implantation (Experimental): Hydrophilic acrylic lens implantation through a micro-incision phacoemulsification and cataract surgery (MICS)
  Interventions: Procedure: IOL implantation; Device: IOL Implantation

INTERVENTIONS:
Procedure: IOL implantation — Micro-incision phacoemulsification cataract surgery (C-MICS) and IOL implantation with 1.8mm cartridge tip insertion technique.
Device: IOL Implantation — Micro-incision phacoemulsification cataract surgery (B-MICS) and IOL implantation with 1.4mm wound-assist insertion technique.

SUMMARY:
The objective of this study is to evaluate clinical outcomes following sub-2 mm micro-incision cataract surgery (MICS) and intraocular lens (IOL) implantation. This study is evaluated in two Phases

* V4 (6M) endpoint: primary analysis
* V5 (12M) and V6 (34M): EPCO score and Nd Yag incidence analysis

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have clear intraocular media other than cataract in the study eye.
* Subjects must have a clinically documented diagnosis of age-related cataract that is considered amenable to treatment with micro-incision phacoemulsification cataract extraction in the study eye.

Exclusion Criteria:

* Subjects with ocular malformation in the study eye.
* Subjects who have had previous surgery in the study eye.
* Subjects with uncontrolled glaucoma in either eye.
* Subjects with any anterior segment pathology for which micro-incision phacoemulsification cataract surgery would be contraindicated
* Subjects using medications known to potentially complicate cataract surgery.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-11-08 (Actual); Primary Completion 2015-06-16 (Actual); Study Completion 2015-06-16 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 6 months
  Corrected distance visual acuity (CDVA)

SECONDARY OUTCOMES:
Incision size | 6 Months
  Incision size before and after implantation
Refraction | 6 Months
  Manifest refraction spherical equivalent. Accuracy to target refraction
Visual Acuity | 6 Months
  Uncorrected distance visual acuity (UDVA)
EPCO | 24 Months
  3 mm evaluation of posterior capsule opacification (EPCO) score
Lens decentration | 6 Months
Laser capsulotomy | 24 Months
  Removal of post-surgical, posterior capsular opacification (PCO)

CONTACTS AND LOCATIONS:
Locations (1):
- Bausch & Lomb, Labège, France